CLINICAL TRIAL: NCT06828887
Title: Multicenter,Randomized,Double-blind,Placebo,Parallel-controlled,Dose-Finding Clinical Trial to Evaluate the Efficacy and Safety of LV232 Capsules in the Treatment of Major Depressive Disorder (MDD)
Brief Title: Dose-Finding Clinical Trial to Evaluate the Efficacy and Safety of LV232 Capsules in the Treatment of MDD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vigonvita Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LV232-MDD-II-01
Record Dates: First submitted 2025-02-10; First posted 2025-02-17 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-02

CONDITIONS: MDD
MeSH Terms: interventions — Population Groups; Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Triple (ParticipantCare ProviderInvestigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- LV232 capsules (Experimental): Capsule, 40 mg or 60 mg, administered orally once daily for 8 consecutive weeks
  Interventions: Drug: LV232 40mg; Drug: LV232 60mg
- Escitalopram (Active Comparator): Tablet, 10 mg , administered orally once daily for 8 consecutive weeks
  Interventions: Drug: Escitalopram
- Placebo (Placebo Comparator): Capsule/Tablet, administered orally once daily for 8 consecutive weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LV232 40mg — LV232 capsules 2 capsules (20 mg/capsule) + LV232 capsule placebo 1 capsule + escitalopram oxalate tablet placebo 1 tablet
  Other Names: Low-dose group
  Arms: LV232 capsules
Drug: LV232 60mg — LV232 capsules 3 capsules (20 mg/capsule) + escitalopram oxalate tablet placebo 1 tablet
  Other Names: High-dose group
  Arms: LV232 capsules
Drug: Escitalopram — LV232 capsule placebo 3 capsule + escitalopram oxalate tablet 1 tablet
  Other Names: Active Comparator
  Arms: Escitalopram
Drug: Placebo — LV232 capsule placebo 3 capsule + escitalopram oxalate tablet placebo 1 tablet
  Other Names: Placebo Comparator,
  Arms: Placebo

SUMMARY:
This multicenter, randomized, double-blind, placebo-controlled, parallel-group, dose-finding Phase II clinical trial aimed to determine the optimal dose of LV232 capsules for treating MDD, evaluate preliminary efficacy and safety, and provide a basis for Phase III trial design and dosing regimen determination.

DETAILED DESCRIPTION:
This study adopts a multicenter, randomized, double-blind, placebo- and active-controlled parallel-group clinical trial design, aiming to evaluate the efficacy and safety of LV232 capsules ( 40 mg, and 60 mg, once daily) in patients with major depressive disorder (MDD).

The trial plans to enroll 400 subjects, stratified by first episode or recurrence of the disease. Participants will be randomized in a 1:1:1:1 ratio into five groups: LV232 capsules 40 mg, 60 mg, placebo, and active control, with 100 subjects in each group. The treatment will be administered once daily for 8 consecutive weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the purpose, content, and potential adverse reactions of this trial, voluntarily participate in the clinical trial and sign a written informed consent form, able to complete the entire trial process as required and comply with the trial regulations;
2. Gender unrestricted, at screening: 18 years old ≤ age ≤ 65 years old;
3. Meet the DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, 5th Edition) diagnostic criteria for depression according to the Mini International Neuropsychiatric Interview (M.I.N.I. 7.0.2), currently experiencing a single or multiple episodes;
4. For first-episode patients, the duration of the current depressive episode must be ≥3 months; for recurrent patients, the duration of the current depressive episode must be ≥1 month (each month is counted as 30 days, the same applies below);
5. During the screening and baseline periods, the total score on the Montgomery-Asberg Depression Rating Scale (MADRS) must be ≥26, and the Clinical Global Impression-Severity (CGI-S) score must be ≥4;
6. At screening and baseline visits, the score on the first item (depressed mood) of the HAMD-17 scale must be ≥2;
7. Female or male subjects of childbearing potential agree and commit to using effective contraception from the signing of the informed consent form until 3 months after the last administration of the trial drug.

Exclusion Criteria:

1. Treatment-resistant depression (failure to respond to an adequate dose and duration of treatment, at least 8 weeks, with two antidepressants of different mechanisms) or failure to respond to an adequate dose and duration of treatment with escitalopram oxalate;
2. Meeting the diagnostic criteria for other mental disorders as per DSM-5 (such as schizophrenia spectrum and other psychotic disorders, bipolar and related disorders, generalized anxiety disorder, obsessive-compulsive and related disorders, somatic symptom and related disorders, etc.);
3. Meeting the DSM-5 criteria for substance use disorder;
4. Organic mental disorders, such as depression caused by hypothyroidism;
5. Depression induced by psychoactive substances or non-addictive substances;
6. Presence of depressive symptoms due to other diseases or other types of mental disorders;
7. A reduction of ≥25% in the MADRS score at baseline compared to the screening period;
8. Assessed by the Columbia Suicide Severity Rating Scale (C-SSRS) and judged by the investigator to be at risk of suicide, or having suicidal behavior within the 6 months prior to screening;
9. Presence of severe physical illnesses deemed by the investigator as grounds for exclusion, such as uncontrolled hypertension or severe unstable cardiovascular diseases, severe liver diseases, kidney diseases, blood diseases, endocrine diseases, neurological diseases, etc.;
10. Diseases affecting oral drug absorption, such as active bowel disease, partial or complete intestinal obstruction, chronic diarrhea, etc.;
11. Active malignancy or a history of malignancy within 5 years prior to screening (except for completely resected and cured squamous cell carcinoma, cervical carcinoma in situ, etc.);
12. History of increased intraocular pressure or narrow-angle glaucoma;
13. Individuals with allergic constitution, such as those allergic to two or more drugs or known to be allergic to escitalopram oxalate;
14. Use of drugs that alter the activity of liver enzymes (CYP2C19 and CYP2D6) within 4 weeks (or 5 half-lives, whichever is longer) prior to randomization (see Appendix 2);
15. Previous treatment with vagus nerve stimulation (VNS) and deep brain stimulation (DBS), or modified electroconvulsive therapy (MECT) within 3 months prior to randomization, or systematic psychotherapy (interpersonal therapy, dynamic therapy, cognitive behavioral therapy), transcranial magnetic stimulation (TMS), and light therapy within 1 month prior to randomization, or judged by the investigator to currently require such treatments;
16. Systematic antidepressant treatment within 2 weeks prior to randomization (not less than 30 days for fluoxetine), or discontinuation of psychotropic drugs for less than 5 half-lives prior to randomization (except for stable doses of sleep aids received within 4 weeks prior to randomization, including benzodiazepines (limited to estazolam, alprazolam, and oxazepam) and non-benzodiazepines);
17. Use of monoamine oxidase inhibitors such as phenelzine, isocarboxazid, tranylcypromine, etc., and linezolid, methylene blue, etc., within 2 weeks prior to randomization;
18. Second or third-degree atrioventricular block, long QT syndrome, or QTcF > 450 ms (male)/460 ms (female) on 12-lead ECG at screening;
19. Discontinuation of drugs that prolong the QT interval (such as levofloxacin, fluconazole, ondansetron, amiodarone, metronidazole, erythromycin, and haloperidol, etc.) or drugs that may cause QT interval prolongation and induce torsade de pointes (TdP) for less than 5 half-lives at randomization;
20. ALT or AST above 2 times the upper limit of normal; creatinine above 1.5 times the upper limit of normal; 2 or more abnormal indicators in thyroid function tests (TSH, FT3, FT4, TT3, or TT4 below 0.9 times the lower limit of normal or above 1.1 times the upper limit of normal) at screening;
21. Positive for Treponema pallidum antibody and HIV antibody at screening;
22. Substance abuse (including alcohol, drugs, and other psychoactive substances) within 3 months prior to screening;
23. Female subjects who are breastfeeding or have a positive pregnancy test at screening or during the trial;
24. Participation in any interventional clinical trial and use of investigational drugs or medical devices within 3 months prior to screening, or currently participating in other clinical trials;
25. Other factors deemed by the investigator as unsuitable for participation in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Montgomery Asperger Depression Scale (MADRS) score at the end of treatment (week 8) | Baseline and week 8
  The MADRS is a clinician-rated scale used to evaluate depressive symptoms over the preceding week. Participants are assessed on 10 items-including feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating, and lack of interest-each scored on a 7-point scale (0 = no symptoms, 6 = maximum severity). The total score ranges from 0 to 60, with higher scores indicating greater depression severity. A negative change in score signifies improvement.
  Change = (Week 8 post-dose score - baseline week 0 score). at the end of treatment (week 8)

SECONDARY OUTCOMES:
Change from baseline in Hamilton Depression Scale (HAMD-17) at week 8 | Baseline, week 8
  The HAMD-17 is a 17-item, clinician-rated scale that assesses depressive symptoms. The HAMD-17 consists of 17 symptoms, each of which is rated from 0 to 2 or 0 to 4, where 0 is none/absent. The HAMD-17 total score is calculated as the sum of the 17 individual symptom scores; the total score can range from 0 to 52. Higher HAMD-17 scores indicate more severe depression.
  Change = (Week 8 post-dose score - baseline week 0 score).
Change from baseline in Hamilton Anxiety Inventory (HAMA) scores at week 8 | Baseline, week 8
  The HAMA is used as a rating measure of anxiety severity. The scale consists of 14 items. Each item is rated on a scale of 0 to 4. The HAMA total score is the sum of the 14 items and the score ranges from 0 to 56, 0 is considered the best outcome.
  Change = (Week 8 post-dose score - baseline week 0 score).
Change from baseline in CGI-S score at week 8 | Baseline and week 8
  The CGI-S is a 7-point scale that requires the clinician to rate the severity of the participant's illness at the time of assessment. The CGI-S will provide an overall clinician-determined summary measure that takes into account all available information including knowledge of the participant's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the participant's ability to function.
  Change = (Week 8 post-dose score - baseline week 0 score).
CGI-I score at week 8 | Baseline, week 8
  The CGI-I assesses the subject's improvement (or worsening). The rater is required to assess the subject's condition relative to baseline* on a 7-point scale. In all cases, the assessment should be made independent of whether the rater believes the improvement is study medication-related or not.
Change from baseline in PHQ-9 score at week 8 | Baseline, week 8
  The PHQ-9 scale consists of 9 items, each corresponding to a core symptom of depression, including depressed mood, loss of interest, sleep disturbances, fatigue, changes in appetite, feelings of guilt, difficulty concentrating, psychomotor retardation or agitation, and suicidal thoughts. Patients are required to rate each item based on their experiences over the past two weeks, with scores ranging from 0 (not at all) to 3 (nearly every day). The total score ranges from 0 to 27, with higher scores indicating more severe depressive symptoms.
Change from baseline in PDQ-D5 score at week 8 | Baseline, week 8
  The PDQ-D5 is used to assess cognitive symptoms, describing potential issues that participants may experience with memory, attention, or concentration. Based on their experiences over the past 7 days, participants select the most appropriate option for each item. The scale consists of 5 items, each with 5 response options (scored 0-4). The total score ranges from 0 to 20, with higher scores indicating more severe cognitive symptoms.
Change from baseline in DSST score at week 8 | Baseline and week 8
  The DSST (Digit Symbol Substitution Test) is used to assess processing speed, attention, and visuomotor coordination. Based on a digit-symbol coding key where each number 1-9 corresponds to a unique symbol, participants match as many symbols to their corresponding numbers as possible within 90 seconds. Higher scores indicate better cognitive function.
Change from baseline in SHAPPS score at week 8 | Baseline and week 8
  The SHAPS (Snaith-Hamilton Pleasure Scale) consists of 14 items assessing hedonic responses to common daily life situations, including but not limited to eating, hobbies/recreational activities, and other typical sources of pleasure.
SMQD score at week 8 | Baseline and week 8
  The Somatic Symptoms Questionnaire for Mental Disorders (SQMD) is a self-rated assessment tool primarily designed to evaluate the severity of common somatic symptoms associated with psychiatric disorders-including depressive disorders, bipolar disorders, anxiety disorders, and somatic symptom disorders-over the past week.
MARS score at week 8 | week 8
  The Medication Satisfaction Rating Scale (MSRS) is a self-rated questionnaire designed to assess patients' satisfaction levels with their current medication regimen.
Change from baseline in ASEX score at week 8 | Baseline and week 8
  The Arizona Sexual Experience Scale (ASEX) is a 5-item rating scale where each item is scored from 1 (hyperfunction) to 6 (hypofunction), with gender-specific versions (male and female) tailored to the assessed individual.
Change from baseline in C-SSRS score at week 8 | Baseline and week 8
  The Columbia Suicide Severity Rating Scale (C-SSRS) is a standardized clinical instrument specifically designed for the assessment of suicide risk.
Incidence of adverse events (AE) | Throughout the study period
  The AEs will be assessed according to the National Cancer Institute (NCI) CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Li Huafang, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center Ethics Committee, Shanghai, China

IPD SHARING:
Plan to Share IPD: No